CLINICAL TRIAL: NCT03916978
Title: Investigating Reactivation of Ovarian Function Following Autologous PRP Intra-ovarian Infusion in Menopausal Women
Brief Title: Autologous PRP Intra Ovarian Infusion to Restore Ovarian Function in Menopausal Women
Acronym: PRP
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Genesis Athens Clinic (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRP - Menopausal women
Record Dates: First submitted 2017-10-25; First posted 2019-04-16 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Infertility, Female; Anovulatory Infertility; Menopause; Amenorrhea
Keywords: Ovarian rejuvenation; Ovarian reactivation; ovulation
MeSH Terms: conditions — Infertility, Female; Amenorrhea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants receiving PRP treatment (Experimental): Menopausal women minimum 45 years of age, receiving ovarian PRP treatment.
  Interventions: Biological: Autologous PRP intra ovarian infusion
- Control Group: Participants receiving Platelet Free Plasma (Placebo Comparator): Women in menopause, 45-55 years old, treated with autologous PFP intra ovarian infusion.
  Interventions: Biological: Autologous PFP intra ovarian infusion

INTERVENTIONS:
Biological: Autologous PRP intra ovarian infusion — Autologous PRP intra ovarian infusion
  Arms: Participants receiving PRP treatment
Biological: Autologous PFP intra ovarian infusion — Autologous PFP intra ovarian infusion
  Arms: Control Group: Participants receiving Platelet Free Plasma

SUMMARY:
Autologous PRP intra ovarian infusion may restore ovarian function, may promote folliculogenesis and may improve hormonal profile of women in menopause.

DETAILED DESCRIPTION:
This triple-blind Randomized Controlled Trial (RCT) aims to investigate the effectiveness of autologous PRP intra ovarian infusion on reactivating ovarian functionality and on promoting folliculogenesis in regard to menopausal women. PRP is blood plasma prepared from fresh whole blood that has been enriched with platelets. It is collected from peripheral veins and contains several growth factors such as vascular endothelial growth factor (VEGF), epidermal growth factor (EGF), platelet derived growth factor (PDGF), transforming growth factor (TGF) and other cytokines all of which stimulate tissue proliferation and growth. PRP has been employed in several medical conditions in Orthopedics, Dermatology, and Ophthalmology for wound healing. It's efficacy in ovarian rejuvenation and reactivation and endometrial regeneration has not been fully elucidated. This study aims to investigate the effect of autologous PRP intra ovarian infusion on restoring ovarian tissue functionality in menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45-55 years old
* Amenorrhea for at least 12 months
* Discontinuation of any complementary/adjuvant treatment including hormone replacement, acupuncture, and botanotherapy, for at least three months prior to recruitment.
* Willing to comply with study requirements

Exclusion Criteria:

* Any pathological disorder related to reproductive system anatomy
* Previous POI diagnosis
* Abnormal karyotype
* Endometriosis
* Adenomyosis
* Fibroids and adhesions
* Infections in reproductive system
* Current or previous diagnosis of reproductive system cancer
* History of familiar cancer in reproductive system
* Severe male factor infertility
* Prior referral for PGT
* Ovarian inaccessibility
* Endocrinological disorders (Hypothalamus-Pituitary disorders, thyroid dysfunction, diabetes mellitus, metabolic syndrome)
* BMI>30 kg/m2 or BMI<18.5 kg/m2
* Systematic autoimmune disorders

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2019-05-21 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Restoration of menstrual cycle | Three months
  Menstrual cycle restoration
Serum FSH levels | Follow-up period of three months entailing monthly evaluation
  Serum FSH levels evaluated monthly for three consecutive months.

SECONDARY OUTCOMES:
Serum AMH levels | Follow-up period of three months entailing monthly evaluation
  Serum AMH levels evaluated monthly for three consecutive months.
Serum estradiol levels | Follow-up period of three months entailing monthly evaluation
  Serum estradiol levels evaluated monthly for three consecutive months.
Serum LH levels | Follow-up period of three months entailing monthly evaluation
  Serum LH levels evaluated monthly for three consecutive months.
Serum progesterone levels | Follow-up period of three months entailing monthly evaluation
  Serum progesterone levels evaluated monthly for three consecutive months.
Antral Follicle Count | Follow-up period of three months entailing monthly evaluation
  AFC evaluated monthly, on day 2 of the menstrual cycle, for three consecutive months.

CONTACTS AND LOCATIONS:
Overall Officials: Agni Pantou, MD, Principal Investigator — Centre of Human Reproduction, Genesis Athens Clinic
Locations (1):
- Genesis AC, Athens, Greece